CLINICAL TRIAL: NCT02606435
Title: Safety and Efficacy of Thrombus Aspiration in Patients With ST-segment Elevation Myocardial Infarction (STEMI)
Brief Title: Thrombus Aspiration in Patients With STEMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, sunddong, Principal Investigator, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEED
Record Dates: First submitted 2015-11-11; First posted 2015-11-17 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: ST-segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- thrombus aspiration with PCI (Experimental): patient will receive manual thrombus aspiration with percutaneous coronary intervention (PCI)
  Interventions: Procedure: percutaneous coronary intervention (PCI); Device: thrombus aspiration
- PCI alone (Active Comparator): patients will receive percutaneous coronary intervention (PCI) alone including stent implantation
  Interventions: Procedure: percutaneous coronary intervention (PCI)

INTERVENTIONS:
Procedure: percutaneous coronary intervention (PCI) — percutaneous coronary intervention (PCI) by stent implantation
  Other Names: primary percutaneous coronary intervention (PCI)
Device: thrombus aspiration — thrombus aspiration with export catheter
  Other Names: export catheter
  Arms: thrombus aspiration with PCI

SUMMARY:
This is a prospective, randomized study with blinded outcome assessment, comparing routine manual thrombus aspiration with no aspiration in patients with acute ST-segment elevation myocardial infarction (STEMI) underwent percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
This is a prospective, randomized study with blinded outcome assessment, comparing routine manual thrombus aspiration with no aspiration in patients with acute ST-segment elevation myocardial infarction (STEMI) underwent percutaneous coronary intervention (PCI). Patients who are diagnosed as STEMI and referred for PCI will be enrolled. They will be randomized 1:1 to either manual thrombus aspiration with PCI group or PCI alone group.The primary outcome is the composite of cardiovascular death, recurrent myocardial infarction (MI), cardiogenic shock, stroke, new or worsening NYHA class IV heart failure during 1 year follow-up. The secondary efficacy outcome are stent thrombosis, target vessel revascularization, left ventricular function and quality of life during 1 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80;
* Diagnosed as STEMI for presenting symptoms or definite ECG and myocardial markers changes;
* Patients presenting with definite ECG changes indicating STEMI: ST elevation of 0.1 mV in 2 contiguous limb leads or ≥0.2 mV in 2 contiguous precordial leads;
* Referred for PCI for presenting symptoms, and the coronary angiogram (CAG) shows that the initial TIMI thrombus grade ≥2;
* Informed consent.

Exclusion Criteria:

* Previous history of myocardiopathy, valvular heart disease or severe heart failure;
* Severe hepatic or renal dysfunction;
* Life expectancy less than 1 year;
* Prior PCI or CABG;
* Contraindications of using anticoagulation or antiplatelet drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | 1 year
  number of participants with cardiovascular death, recurrent myocardial infarction (MI), cardiogenic shock, stroke, new or worsening NYHA class IV heart failure

SECONDARY OUTCOMES:
Number of participants with stent thrombosis | 1 year
  number of participants with stent thrombosis
Number of participants with target vessel revascularization | 1 year
  number of participants with target vessel revascularization
left ventricular function | 1 year
  left ventricular ejection fraction evaluated by ultrasound
Seattle Angina Questionnaire scores | 1 year
  Seattle Angina Questionnaire scores
6-minute walk distance (6MWD) | 1 year
  6-minute walk distance (6MWD)

CONTACTS AND LOCATIONS:
Overall Officials: Dongdong Sun, M.D.,Ph.D., Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China